CLINICAL TRIAL: NCT03997916
Title: A Validation Investigation of the Accuracy of the Belun Ring, an Innovative Single-channel Four-signal Pulse Oximetry, in Patients Referred to Sleep Lab for Assessment of Obstructive Sleep Apnea
Brief Title: Belun Ring Validation Study for Assessment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Belun Technology Company Limited (Other)
Responsible Party: Principal Investigator, Eric Yeh, MD, Fellow in Sleep Medicine, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY20181042
Record Dates: First submitted 2019-06-23; First posted 2019-06-25 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Belun Ring; pulse oximeter; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participant (Other): All patients scheduled for attended overnight in-lab polysomnography (PSG), also known as sleep study, in our 2 sleep labs will undergo PSG testing. On the same night of the PSG testing, these same patients will also wear the Belun Ring device. After the study, we will compare results of the Belun Ring device vis-à-vis with the results of the PSG on the same patient. There will be no separate arm to test a different device.
  Interventions: Device: Belun Ring; Diagnostic Test: PSG

INTERVENTIONS:
Device: Belun Ring — All patients scheduled for attended overnight in-lab polysomnography (PSG) in our 2 sleep labs will undergo PSG testing. On the same night of the PSG testing, these same patients will also wear the Belun Ring device. After the study, we will compare results of the Belun Ring device vis-à-vis with the results of the PSG on the same patient.
Diagnostic Test: PSG — All patients scheduled for attended overnight in-lab polysomnography (PSG) in our 2 sleep labs will undergo PSG testing. On the same night of the PSG testing, these same patients will also wear the Belun Ring device. After the study, we will compare results of the Belun Ring device vis-à-vis with the results of the PSG on the same patient.

SUMMARY:
This study aims to determine the overall accuracy, sensitivity, and specificity of the Belun Ring device in evaluating obstructive sleep apnea by comparing the device to the attended overnight in-lab polysomnography which is the gold standard for diagnosis of obstructive sleep apnea. Our hypothesis is that the Belun-Ring, a type 4 portable monitoring device, is overall sensitive and specific for evaluation of obstructive sleep apnea when compared to the attended overnight in-lab polysomnography.

DETAILED DESCRIPTION:
This study will include all patients who are scheduled to do an attended overnight in-lab polysomnography in 2 sleep labs owned by University Hospitals Cleveland Medical Center. These patients will receive email recruitment forms 2 weeks prior their scheduled polysomnography. Whether they are interested or not, patients are supposed to call or email the study's central contact person. Both phone number and email address of the central contact person are noted in the email recruitment form. For those patients who did not make any contact with the study's central contact person, they will be screened for eligibility by sub-investigators through chart review. List of eligible patients will be sent to the central contact backup person who is basically in-charge of making phone calls to the patients. This person will further confirm patients' eligibility over the phone and ask if they are interested. If a patient is interested, the central contact backup person will inform the sub-investigators who, in turn, will assign a unique patient identifier to the interested subject and inform the sleep lab contact person. The sleep lab contact person will, in turn, inform the sleep technicians on-call ahead of time about the list of interested subjects. On the night of the polysomnography testing of the interested subject, the latter will receive questionnaires and written informed consent form related to the study which will be explained by the sleep technician. After the subject had completed and signed the questionnaires and written informed consent form respectively, the sleep technician will apply the Belun Ring device on the patient as well as the electrodes and sensors included in a routine polysomnography. The following day, data from Belun Ring device will be uploaded to the laptop while another sleep technician will read the polysomnography. Sub-investigators will enter the data from the questionnaires, Belun Ring device, and polysomnography in the secured University Hospitals Redcap (UHRedcap). Once the target number of subjects are reached, all data will be sent to statistician for analysis.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients age 18-80 years old scheduled for overnight in-lab sleep study
* Provision of signed and dated written informed consent form

Exclusion Criteria:

* Recent hospitalization in the past 30 days
* Patients on home oxygen, non-invasive ventilator, diaphragmatic pacing, or any form of nerve stimulator
* Patients with pacemaker, defibrillator, left ventricular assist device (LVAD), or status post cardiac transplantation
* Patients with baseline heart rate under 50 bpm or over 100 bpm during last clinic visit or prior to study at the sleep lab
* Patients with unstable cardiopulmonary status judged to be unsafe for sleep study by the sleep technician and/or the on-call sleep physician in the sleep lab on the night of the study
* Patients who are unable to complete the required study
* Patients involved in another investigational study
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Yeh, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Ambrose Chiang, MD, Study Director — University Hospitals Cleveland Medical Center; Kingman Strohl, MD, Study Director — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - Residence Inn Marriott, Beachwood, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeh E, Wong E, Tsai CW, Gu W, Chen PL, Leung L, Wu IC, Strohl KP, Folz RJ, Yar W, Chiang AA. Detection of obstructive sleep apnea using Belun Sleep Platform wearable with neural network-based algorithm and its combined use with STOP-Bang questionnaire. PLoS One. 2021 Oct 11;16(10):e0258040. doi: 10.1371/journal.pone.0258040. eCollection 2021. PMID 34634070
- Available data/document: Individual Participant Data Set — http://redcap.uhhospitals.org/redcap

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 336 subjects were screened, 130 subjects did not meet eligibility criteria. Out of the 206 subjects who were eligible, 93 refused to participate.
  Total of 113 subjects completed informed consent process and enrolled in the study.
Groups:
- Participant: All patients scheduled for attended overnight in-lab polysomnography (PSG), also known as sleep study, in our 2 sleep labs will undergo PSG testing. On the same night of the PSG testing, these same patients will also wear the Belun Ring device. After the study, we will compare results of the Belun Ring device with the results of the PSG on the same patient. There will be no separate arm to test a different device.
  Belun Ring: All patients scheduled for attended overnight in-lab polysomnography (PSG) in our 2 sleep labs will undergo PSG testing. On the same night of the PSG testing, these same patients will also wear the Belun Ring device. After the study, we will compare results of the Belun Ring device with the results of the PSG on the same patient.
  PSG: All patients scheduled for attended overnight in-lab polysomnography (PSG) in our 2 sleep labs will undergo PSG testing. On the same night of the PSG testing, these same patients will also wear the Belun Ring device. After the study, we will compare results of the Belun Ring device with the results of the PSG on the same patient.
Period: Overall Study
Arm/Group | Participant
Started | 113
Completed | 78
Not Completed | 35
Not completed — Protocol Violation | 35

BASELINE CHARACTERISTICS:
Population: subjects that are eligible and willing to be consented to participate in the study and whose length of data recording is sufficient for Belun Ring Analysis
Arm/Group | Participant
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 41
  White | 4
  More than one race | 0
  Unknown or Not Reported | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 36.1 (10.1)
STOP-Bang [Mean (Standard Deviation); unit: scores on a scale] — S.T.O.P. - B.A.N.G. is an acronym, which stands for Snoring, Tiredness, Observed apnea, blood Pressure, Body mass index, Age, Neck circumference and Gender. This questionnaire was specifically developed to meet the need for a reliable, concise, and easy-to-use screening tool. It consists of eight dichotomous (yes/no) items related to the clinical features of sleep apnea. The total score ranges from 0 to 8. With 0 being low risk and 8 being high risk for obstructive sleep apnea.
  scores on a scale | 3.9 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Performance (Mean With 95% CI) of bAHI at PSG--AHI Cutoffs of 5, 15 and 30 (Accuracy)
Description: Comparing the accuracy, sensitivity, specificity of Belun Ring Device versus gold standard Polysomnography for Obstructive Sleep Apnea
Time Frame: Same night when both testing were done on the same subject
Measure: Number (95% Confidence Interval); unit: proportion of events
Groups:
- Belun Ring Study Participants: Subjects that are eligible, willing to consent and completed the study with sufficient data for analysis
Arm/Group | Belun Ring Study Participants
Number analyzed (Participants) | 78
proportion of events
  AHI cut off of 5 | 0.564 [0.447 to 0.676]
  AHI cut off of 15 | 0.808 [0.703 to 0.888]
  AHI cut off of 30 | 0.910 [0.824 to 0.963]

2. Primary Outcome: Sensitivity
Description: as for outcome 1
Time Frame: Same night when both testing were done on the same subject
Measure: Number (95% Confidence Interval); unit: proportion of events
Arm/Group | Belun Ring Study Participants
Number analyzed (Participants) | 78
proportion of events
  AHI cut off at 5 | 1.000 [0.918 to 1.000]
  AHI cut off at 15 | 0.931 [0.772 to 0.992]
  AHI cut off at 30 | 0.714 [0.419 to 0.916]

3. Primary Outcome: Specificity
Description: as for outcome 1
Time Frame: Same night when both testing were done on the same subject
Measure: Number (95% Confidence Interval); unit: proportion of events
Arm/Group | Belun Ring Study Participants
Number analyzed (Participants) | 78
proportion of events
  AHI cut off of 5 | 0.029 [0.001 to 0.149]
  AHI cut off of 15 | 0.735 [0.589 to 0.850]
  AHI cut off of 30 | 0.953 [0.869 to 0.990]

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Belun Ring Device: Affected / at Risk (%)
Arm/Group | Belun Ring Device
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT03997916/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT03997916/ICF_001.pdf